CLINICAL TRIAL: NCT03130413
Title: Comparing the Effectiveness Between Air-Q Intubating Laryngeal Airway and Ambu® AuraGain™ Laryngeal Mask for Controlled Ventilation in Paediatric Patients: A Randomized Controlled Trial.
Brief Title: Comparing Between Air-Q Intubating Laryngeal Airway and Ambu® AuraGain™
Acronym: Nira
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Ambu A/S (Industry)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/15110476
Record Dates: First submitted 2017-04-02; First posted 2017-04-26 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: General Anaesthesia
Keywords: Ambu Aura Gain; Air-Q intubating laryngeal airway; Paediatric surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambu Aura Gain (Experimental): Ambu Aura Gain supraglottic airway size 2 or 2.5 will be inserted once patients are paralyzed
  Interventions: Device: Ambu Aura Gain supraglottic airway
- Air-Q (Active Comparator): Air-Q supraglottic airway size 1.5 and 2.0will be inserted once the patients are paralyzed
  Interventions: Device: Air-Q supraglottic airway

INTERVENTIONS:
Device: Ambu Aura Gain supraglottic airway — Anesthesia is induced with sevoflurane in oxygen. The anesthesia plane is gradually deepened by increasing the inspired concentration of sevoflurane (2-8%) till the loss of eyelash reflex. After intravenous (IV) cannula is inserted and intravenous fentanyl 1mcg/kg and rocuronium 0.6mg/kg are administered. Use of neuromuscular blocking agent is to minimize the risk of reflex activation of the airway. After 3 minutes, the appropriate size (depending upon body weight) of Ambu Aura Gain is lubricated with water soluble lubricant (KY jelly) is inserted by investigator based on manufacturer recommendation with the patient's head in neutral position. The cuff then is inflated to an intra-cuff pressure of 40 cm H20, measured using a digital cuff pressure monitor.
  Arms: Ambu Aura Gain
Device: Air-Q supraglottic airway — Anesthesia is induced with sevoflurane in oxygen. The anesthesia plane is gradually deepened by increasing the inspired concentration of sevoflurane (2-8%) till the loss of eyelash reflex. After intravenous (IV) cannula is inserted and intravenous fentanyl 1mcg/kg and rocuronium 0.6mg/kg are administered. Use of neuromuscular blocking agent is to minimize the risk of reflex activation of the airway. After 3 minutes, the appropriate size (depending upon body weight) of Air-Q supraglottic airway is lubricated with water soluble lubricant (KY jelly) is inserted by investigator based on manufacturer recommendation with the patient's head in neutral position. The cuff then is inflated to an intra-cuff pressure of 40 cm H20, measured using a digital cuff pressure monitor.
  Arms: Air-Q

SUMMARY:
The aim of this randomized study is conducted is to evaluate the performance and safety of air-Q intubating laryngeal airway as primary airway device in various short surgical procedure in children compared to Ambu® AuraGain™ Laryngeal Mask. Current Supraglottic airway devices (SADs) available in are classic LMA (cLMA), proseal LMA (pLMA), supreme LMA (sLMA) and the newer is Ambu® AuraGain™laryngeal mask. As variety of newer SADs for children have emerged since their introduction in clinical practice, hope the outcomes of this study it help advancing our knowledge and acumen in selecting appropriate devices for paediatric population.

DETAILED DESCRIPTION:
JUSTIFICATION OF STUDY

In view of no clinical data is available evaluating the clinical performance and safety of air-Q and Ambu® AuraGain™ in children, therefore this prospective and randomized study is conducted. Most of previous randomized studies in term of safety did not compare the hemodynamic stability.Hope the outcomes of this study it help advancing our knowledge and acumen in selecting devices for paediatric population.

RESEARCH HYPOTHESES

1. There is no difference in the ease of insertion (number of attempts and time of insertion) between air-Q and Ambu® Aura Gain™.
2. There is no difference in the oropharyngeal leak pressure (OLP) between air-Q and Ambu® Aura Gain™.
3. There is no difference in hemodynamic changes between air-Q and Ambu® Aura Gain™.
4. There is no difference in the incidence of complications between air-Q and Ambu® Aura Gain™.

METHODOLOGY

This is a prospective, single blinded and randomized controlled trial study will be conducted at Operation Theatre (OT), Hospital University Sains Malaysia (HUSM). involving paediatric patients scheduled for various surgical procedures within 2 hours where supraglottic airway management would be appropriate..

Sample size calculation For objective 1, sample size was calculated using power and sample size software and the data based on previous study by V.Darlong et al (Comparison of air-Q and Ambu Aura-i for controlled ventilation in infants: a randomized controlled trial). In this study, the time for successful insertion for air-Q is 16.53±1.53 and Ambu Aura-I is 14.68±2.83. Considering power of 80% and type error-I α of 5%, the sample size was required is 15 participants in each group. 10% is added for drop out sample. Therefore sample size, n 15 + (0.1x15) = 17 participants for each group.

For objective 2, sample size was calculated using power and sample size software and the data based on previous study by V.Darlong et al (Comparison of air-Q and Ambu Aura-i for controlled ventilation in infants: a randomized controlled trial). In this study, the OLP for air-Q is 20.21±4.62 and Ambu Aura-I is 16.21±5.66. Considering power of 80% and type error-I α of 5%, the sample size was required is 22 participants in each group. 10% is added for drop out sample. Therefore sample size, n 22 + (0.1x22) = 25 participants for each group.

Overall sample size is estimated using objective 2 because of larger sample size. Total sample size is 50 patients.

SAMPLING METHOD Patients are randomly assigned into 2 groups: air-Q (A) and Ambu® AuraGain™ (B) using computer-generated randomization. Sequentially-numbered sealed opaque envelopes containing group allocation as determined by computer-generated sequence, will be opened by a nurse in charge for study device preparation.

RECRUITMENT OF SUBJECT & INFORMED CONSENT SEEKING Paediatric patients who meets the study criteria, their parents will be approached to invite patients participate in this study. Each parent will be given a thorough explanation along with copy of Patient Information Sheet. All questions that the participant's parents have, will be answered to their satisfaction before consent been obtained by signing the consent form.

The study is divided into screening, pre-operative, intra-operative and post-operative period.

1. Screening period After obtaining approval from the Ethics committee, participants will be selected according to inclusion and exclusion criteria during preoperative assessment round. Study procedures will be explained and written consent will be obtained from the participant's parents.
2. Pre-operative period In all participants, a eutectic mixture of local anaesthetic cream (EMLA) will be applied on both hands 30 minutes before transfer to operation theatre. No premedication will be prescribed in the morning of the surgery. All consented participants will be randomized using computer generated randomization into two groups: Group a (air-Q) and group B (Ambu Aura Gain). All demographic data including types and duration of surgery and diagnosis of procedure is recorded.
3. Intra-operative Anaesthesia Technique In operation theatre, all of the participants will be monitored with non-invasive blood pressure (NIBP), pulse oximeter (SpO2), electrocardiogram (ECG) and capnography (EtCO2). Anesthesia is induced with sevoflurane in oxygen. The anesthesia plane is gradually deepened by increasing the inspired concentration of sevoflurane (2-8%) till the loss of eyelash reflex. An intravenous (IV) cannula is inserted and intravenous fentanyl 1mcg/kg and rocuronium 0.6mg/kg are administered. Use of neuromuscular blocking agent is to minimise the risk of reflex activation of the airway. After 3 minutes, the appropriate size (depending upon body weight) of SADs (according to the group allocated based on the sequence of computerized randomization) lubricated with water soluble lubricant (KY jelly) is inserted by the investigator by standard technique as per manufacture's recommendation. Then the cuff is inflated and intracuff pressure is then standardized to 60 cmH20 using a digital cuff pressure monitor. Data and timing are collected by independent observers. To prevent biasedness in conducting the study, the same investigator will insert the device for all participants.

   Haemodynamic parameters such as blood pressure (BP), heart rate (HR), oxygen saturation (SpO2) and end tidal carbon dioxide (EtCO2) is recorded at different interval namely, pre induction, post induction, post insertion, every 2 minutes for 10 minutes and then 5 minutes thereafter until extubation.

   Anesthesia is maintained with sevoflurane (Minimum Alveolar Concentration value of 1.0-1.2) in Oxygen: Air mixture of 50% . Pressure controlled ventilation is set and targeting the minute ventilation to achieve normocarbia (EtCO2 35-40 mmHg). Intra-operative analgesia is supplement by suppository paracetamol 20 mg/kg or diclofenac sodium 1mg/kg.

   Measurement of parameters
   1. Attempts required to successfully insert the device is recorded
   2. A successful insertion is defined as visible chest rise and a square wave trace on the capnograph. Failure of device is labelled where need more than 3 attempts to insert the device or alternative device is inserted or trachea is intubated.
   3. The time from the picking up the device and chest rise with positive pressure ventilation is recorded as time to insert.
   4. Oropharyngeal leak pressure (OLP) is recorded by observing the peak airway pressure at which audible leak occurred at the first time when fresh gas flow delivered at 3 litre/min and the expiratory valve is completely closed. For safety, OLP is not allowed to exceed >40 cmH20.
   5. Failure of device is also labelled if any intra-operative device repositioning or replacement of the device due to excessive air leak or airway obstruction as evidenced by an obstructive pattern on the capnograph leading to desaturation.
4. Post-Operative At the end of surgery, sevoflurane is turned off and 100% oxygen is administered. Muscle relaxant is reversed by neostigmine (50 mcg/kg) and glycopyrrolate (10 mcg/kg). With adequate tidal volume and respiratory rate, oropharyngeal suctioning is done and the device is removed. On removal of the device, any presence of blood stain or tongue-lip-dental trauma is recorded. In the post-operative period, the participant is observed for any complications such as airway reflex activation (laryngospasm, bronchospasm or severe cough), oxygen desaturation (spO2 <90%) and vomiting/aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1-6 years
* Weight 10-30kg
* American Society of Anesthesiologist (ASA) physical status class I and II
* Any surgical procedures where supraglottic airway (SGA) management is appropriate
* Duration of procedure within 2hours

Exclusion Criteria:

* Active respiratory infection
* Anticipated and known difficult airway
* Lung disease requiring high airway pressure

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2016-11; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
measure fibreoptic (FO) grade of laryngeal view | 5 minutes after insertion of the device when good tidal volume is achieved
  Flexible fibreoptic scope is use to view anatomical alignment of the device to the larynx, 1cm proximal to the ventilating orifice

SECONDARY OUTCOMES:
oropharyngeal leak pressure (OLP) | 5 minutes after insertion of the device when good tidal volume is achieved
  OLP is recorded by observing the peak airway pressure which audible leak occur at the first time when fresh gas flow delivered at 3 litre/min and the expiratory valve is completely closed
number of attempt | Throughout the insertion process up to 5 minutes post induction
  Measure number of attempts of inserting the devices
Time of insertion | The time from which the device first being hold until successful insertion up to 5 minutes post induction
  Measure the time of successful insertion of the devices
Blood pressure | Time from pre-induction until 5 minutes post insertion
  Documented the blood pressure (BP) is recorded at different time interval
Heart rate | Time from pre-induction until 5 minutes post insertion
  Recorded the heart rate (HR) is recorded at different interval
Oxygen saturation (SpO2) | Time from pre-induction until 5 minutes post insertion
  Oxygen saturation (SpO2) is recorded at different interval
end tidal Carbon dioxide (EtCO2) | Time from pre-induction until 5 minutes post insertion
  The EtCO2 is recorded at different time interval
numbers of adverse effects of the devices as assessed by clinical observation | Throughout the stay in recovery bay within 30 minutes after operation
  Presence of adverse effect of the device postextubation

CONTACTS AND LOCATIONS:
Overall Officials: Rhendra Hardy Mohamad Zaini, MD, Principal Investigator — Universiti of Science Malaysia
Locations (1):
- University of Science Malaysia Hospital, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Darlong V, Biyani G, Baidya DK, Pandey R, Chandralekha, Punj J, Upadhyay AD. Comparison of air-Q and Ambu Aura-i for controlled ventilation in infants: a randomized controlled trial. Paediatr Anaesth. 2015 Aug;25(8):795-800. doi: 10.1111/pan.12663. Epub 2015 Apr 27. PMID 25917434
- [Result] Darlong V, Biyani G, Pandey R, Baidya DK, Punj Ca. Comparison of performance and efficacy of air-Q intubating laryngeal airway and flexible laryngeal mask airway in anesthetized and paralyzed infants and children. Paediatr Anaesth. 2014 Oct;24(10):1066-71. doi: 10.1111/pan.12462. PMID 24961960
- [Result] Jagannathan N, Hajduk J, Sohn L, Huang A, Sawardekar A, Gebhardt ER, Johnson K, De Oliveira GS. A randomised comparison of the Ambu(R) AuraGain and the LMA(R) supreme in infants and children. Anaesthesia. 2016 Feb;71(2):205-12. doi: 10.1111/anae.13330. Epub 2015 Dec 9. PMID 26648173
- [Result] Whyte SD, Cooke E, Malherbe S. Usability and performance characteristics of the pediatric air-Q(R) intubating laryngeal airway. Can J Anaesth. 2013 Jun;60(6):557-63. doi: 10.1007/s12630-013-9918-6. Epub 2013 Mar 22. PMID 23519724